CLINICAL TRIAL: NCT06320366
Title: Testing an Accelerated TMS Protocol for Methamphetamine Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-1044; K24DA058882 (NIH)
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Methamphetamine Use Disorder

STUDY DESIGN:
Intervention Model Description: Sham vs. real Transcranial Magnetic Stimulation (TMS)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant and all study personnel are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sham TMS (Placebo Comparator): Participants have baseline assessments/evaluation, are admitted to the inpatient research unit, randomized via permuted block design to 5 days of sham TMS, and then have weekly study visits for the next 12 weeks.
  Interventions: Device: Sham TMS
- Active TMS (Experimental): Participants have baseline assessments/evaluation, are admitted to the inpatient research unit, randomized via permuted block design to 5 days of active TMS, and then have weekly study visits for the next 12 weeks.
  Interventions: Device: Active TMS

INTERVENTIONS:
Device: Sham TMS — The TMS Cool-B65 A/P coil on its placebo side delivers electrical stimulation to the scalp (e.g., mimicking sensations associated with real stimulation) but does not provide magnetic stimulation to the targeted cortical structure.
  Arms: Sham TMS
Device: Active TMS — The TMS Cool-B65 A/P coil delivers magnetic stimulation to targeted cortical structure.
  Arms: Active TMS

SUMMARY:
The investigators will evaluate the effects of an accelerated Transcranial Magnetic Stimulation (TMS) protocol of the left dorsolateral prefrontal cortex (DLPFC) for moderate to severe methamphetamine use disorder. This is a randomized parallel group design to assess feasibility and safety, evaluate efficacy (use, craving) and identify magnetic resonance imaging (resting state and cue craving) associated with group/outcomes.

DETAILED DESCRIPTION:
In a randomized double-blind parallel-group sham-controlled design (n=20) administer a 5-day accelerated iTBS protocol (40 treatments) to the left dorsolateral prefrontal cortex during a short inpatient stay. Magnetic resonance imaging will be completed pre-post TMS and participants will be followed for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-65 years inclusive;
2. Meets DSM-5 criteria for past-year moderate or severe methamphetamine use disorder;
3. By Timeline Follow Back endorses at least 10 days of methamphetamine use out of the last month;
4. Provides a urine drug screen positive for methamphetamine;
5. Able to provide informed consent;
6. No change in current psychiatric medication regimen, or medication free, for at least 4 weeks prior to study entry;
7. Adequate English proficiency for study consent, and completion of the study instruments.

Exclusion Criteria:

1. Lifetime non-substance-induced psychotic disorders, schizophrenia, schizoaffective disorder or bipolar disorder defined by DSM-5;
2. Current diagnosis of DSM-5 drug use disorder other than stimulant, cannabis or nicotine use disorder;
3. Non-substance-induced manic episode within the past 3 years or major depressive episode in the past year;
4. Current clinically significant neurological disorder or medical illness, including history of seizures, cardiovascular disease/cardiac event, which in the opinion of the study physician would make study participation unsafe;
5. Presence of a clinically significant abnormality on baseline MRI;
6. Inability to have an MRI;
7. Currently breastfeeding, is currently pregnant or lack of use of effective contraception in women of childbearing age, as assessed by urine pregnancy test and self-report (participants will consent to continue effective contraceptives during the study);
8. Active criminal justice involvement (i.e., any unresolved legal problems that could jeopardize continuation or completion of the study);
9. History of head injury with loss of consciousness for more than 15 minutes;
10. Diagnosis of dementia;
11. Prescribed benzodiazepines or anticonvulsants;
12. Currently enrolled in formal substance use disorder treatment;
13. Metal implants or non-removable metal objects above the waist;
14. Lifetime history of prior clinical treatment with TMS;
15. Serious risk of suicide or homicide;
16. Unable/unwilling to follow the study procedures;
17. History of intractable migraine;
18. Assessed to be at risk for alcohol or opioid withdrawal.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Tolerability | 5 days
  Proportion completing at least 20 TMS session - sham vs. active
Study emergent adverse events | 12 weeks
  Incidence of study emergent adverse events - sham vs. active

SECONDARY OUTCOMES:
Weeks of continuous abstinence | 12 weeks
  Number of weeks of continuous methamphetamine abstinence - sham vs. active as measured weekly by urine drug screen.
Days of methamphetamine use | 12 weeks
  Number of days of methamphetamine use - sham vs. active as measured weekly by timeline followback interview.
Time to first methamphetamine use | 12 weeks
  Time from end of TMS treatment to first methamphetamine use by timeline follow back or urine drug screen
Methamphetamine craving | 12 weeks
  Craving as measured on the Stimulant Craving Questionnaire-Brief - sham vs. active. Each item is scored 0-6 (from Strongly Disagree=0 to Strongly Agree=6) with items #4 and #7 reverse scored. The investigators will average all 10 items as the total score, with higher scores indicating greater levels of craving.
Methamphetamine craving on visual analog scale | 12 weeks
  Craving as measured on visual analog scale - sham vs. active. Scored 0 to 100 with 0=no craving and 100=the most craving.
MRI cue craving | Pre- and Post- TMS stimulation in week 1
  Cue craving data will be collected pre- and post-TMS stimulation in week 1
MRI resting state | Pre- and Post- TMS stimulation in week 1
  Resting state data will be collected pre- and post-TMS stimulation in week 1

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.